CLINICAL TRIAL: NCT00319436
Title: Fostering Mothers' Emotionally Responsive Parenting
Brief Title: Stage I Randomized Trial of Mentalization-Based Therapy for Substance Using Mothers of Infants and Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0407026890-B; R01DA017294 (NIH)
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Maternal Substance Use; Child Abuse and Neglect
Keywords: parenting intervention; family intervention; maternal substance abuse; mother-child relations; parent-child relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mentalizing Therapy for Substance Using Mothers (Experimental): This 12 session individual therapy aims to enhance maternal reflective functioning and soften harsh and distorted mental representations about the child. The intervention adopts a developmental progression based on attachment theory, supporting the mother in her parenting role and offering assistance with basic needs. Mothers are encouraged to reflect on their thoughts and feelings and how they affect behavior. The therapist assists mother's thinking about representations of herself as a parent and encourages her to explore opportunities for new understanding of her emotional needs. Therapist and mother explore representations of her child and their relationship in detail in order to understand their meaning and promote more balanced representations and affect regulation. Therapist and mother also explore child's emotional experiences underlying behavior. The goal is to support the mother in becoming more aware of her child's emotional needs.
  Interventions: Behavioral: Mentalizing Therapy for Substance Using Mothers
- Standard Parent Education for Substance Using Mothers (Active Comparator): This 12 session comparison intervention was designed to match the Maternal Mentalizing Therapy on time spent with the counselor and maternal expectations for help with parenting. PE counselors helped mothers get connected to services (e.g. medical and pediatric care, child care and child guidance services, housing assistance, vocational training), solve problems of daily living and make parenting-related decisions. PE mothers also received a pamphlet each week on a parenting topic of their choice. Pamphlets focused on common issues in caring for infants (e.g., soothing a crying baby, managing bedtime routines, and establishing routines ) and toddlers (e.g., helping toddlers dress, managing bedtime battles, managing difficult behavior in public, and setting limits without using punishment). Pamphlets provided behavioral guidance at a 5th grade reading level without reference to underlying mental states or emotional needs.
  Interventions: Behavioral: Standard Parent Education for Substance Using Mothers

INTERVENTIONS:
Behavioral: Mentalizing Therapy for Substance Using Mothers — This 12 session individual therapy aims to enhance maternal reflective functioning and soften harsh and distorted mental representations about the child. The intervention adopts a developmental progression based on attachment theory, supporting the mother in her parenting role and offering assistance with basic needs. Mothers are encouraged to reflect on their thoughts and feelings and how they affect behavior. The therapist assists mother's thinking about representations of herself as a parent and encourages her to explore opportunities for new understanding of her emotional needs. Therapist and mother explore representations of her child and their relationship in detail in order to understand their meaning and promote more balanced representations and affect regulation. Therapist and mother also explore child's emotional experiences underlying behavior. The goal is to support the mother in becoming more aware of her child's emotional needs.
  Arms: Mentalizing Therapy for Substance Using Mothers
Behavioral: Standard Parent Education for Substance Using Mothers — This 12 session comparison was designed to match the experimental intervention on time spent with the counselor and maternal expectations for help with parenting. PE counselors helped mothers get connected to services (e.g. medical and pediatric care, child guidance services, housing assistance, vocational training), solve problems of daily living and make parenting-related decisions. PE mothers also received a pamphlet each week on a parenting topic of their choice. Pamphlets focused on common issues in caring for infants (e.g., soothing a crying baby, managing bedtime routines, and establishing routines ) and toddlers (e.g., helping toddlers dress, managing bedtime battles, managing difficult behavior in public, and setting limits without using punishment). Pamphlets provided behavioral guidance at a 5th grade reading level without reference to underlying mental states or emotional needs.
  Arms: Standard Parent Education for Substance Using Mothers

SUMMARY:
The primary goal of this Stage I therapy development study will be to manualize and test the preliminary efficacy of a parenting intervention for drug dependent mothers that aims to foster their ability to recognize children's emotional needs at different ages and their capacity to be emotionally available to their children.

DETAILED DESCRIPTION:
Mothers who are physically and/or psychologically dependent upon alcohol and drugs are at risk for a wide range of parenting deficits beginning when their children are infants and continuing as their children move through school-age and adolescent years. Behavioral parent training programs for drug dependent mothers have had limited success in improving mother-child relationships or children's psychosocial adjustment. One reason behavioral parenting programs may have had limited success is the lack of attention to emotional aspects of the mother-child relationship, including (1) mothers' recognition of their children's emotional needs and (2) mothers' capacity to respond sensitively to their children's emotional cues. Research on attachment suggests that the emotional quality of the early mother-child relationship has important implications for many developmental capacities, including emotional and behavior regulation in early years, and social competence academic achievement in school-aged and adolescent years. In this Stage I therapy development study, we propose to modify a previously piloted attachment-based group parenting intervention called Emotionally-Responsive Parenting Group or ERP. The goal of the intervention is to improve the mother's capacity to recognize and sensitively respond to her child's emotional cues. In a pre-pilot study (see Preliminary Study 6) we tested the feasibility of conducting the ERP group intervention as an adjunct group treatment for 23 primarily cocaine-dependent mothers in outpatient drug treatment and found that ERP was highly feasible and showed initial promise for improving maternal recognition of emotional cues. In this study, we aim to modify and validate the intervention as an individual therapy for drug dependent mothers of children ages 18 to 36 months in preparation for a Stage II controlled efficacy trial.

More specifically, we will:

1. Develop and modify a 12-session ERP individual therapy for drug dependent mothers enrolled in outpatient drug treatment have custody of a child between 18 and 36 months of age. Fifteen mothers enrolled in outpatient drug treatment will participate in this phase of the ERP manual's development.
2. Develop and implement a therapist training and supervision program for delivery of the ERP manualized treatment. This phase will include the development of ERP adherence and competence rating scales.
3. Conduct a randomized, controlled pilot study to determine the potential feasibility, acceptability, and efficacy of ERP compared with, Parent Education (PE), a 12-week comparison condition in which mothers will attend 12 1-hour parent education sessions conducted by a paraprofessional. Sixty mothers enrolled in outpatient drug treatment who have at least one child between the ages of 18 and 36 months in their custody will participate. Because the intervention will directly target change in maternal psychological representations of parenting, primary outcomes will be (a) maternal 'reflective functioning' (capacity to make inferences about emotional cues, (b) capacity for balanced psychological representations of the child, and (c) knowledge of the child's developmental capacities. The intervention will indirectly target maternal and child behavior and maternal psychosocial adjustment. Secondary outcomes will be: maternal sensitivity to her child's emotional cues, the child's use of the mother as a secure base, and maternal psychiatric distress, daily functioning and substance abuse.
4. Explore the impact of process variables on outcomes, and potential mediator and moderator effects.. Process variables will be: (a) attendance, (b) therapeutic alliance, (c) therapist adherence and competence and (d) use of additional treatment services.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adult women
* history of primary alcohol, cocaine, cannabis, club drug, or heroin abuse or dependence
* caring for a child between 1 and 36 months of age

Exclusion criteria:

* acute suicidality/ homicidality
* severe psychiatric or substance-related symptoms requiring in-patient hospitalization or ambulatory detoxification

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Suchman, Ph.D., Principal Investigator — Yale University
Locations (1):
- The APT Foundation, New Haven, Connecticut, United States

REFERENCES:
- [Background] Suchman N, Mayes L, Conti J, Slade A, Rounsaville B. Rethinking parenting interventions for drug-dependent mothers: from behavior management to fostering emotional bonds. J Subst Abuse Treat. 2004 Oct;27(3):179-85. doi: 10.1016/j.jsat.2004.06.008. PMID 15501370
- [Background] Suchman N, Pajulo M, Decoste C, Mayes L. Parenting Interventions for Drug-Dependent Mothers and Their Young Children: The Case for an Attachment-Based Approach. Fam Relat. 2006 Apr;55(2):211-226. doi: 10.1111/j.1741-3729.2006.00371.x. PMID 17417669
- [Result] Suchman N, Decoste C, Castiglioni N, Legow N, Mayes L. THE MOTHERS AND TODDLERS PROGRAM: Preliminary Findings From an Attachment-Based Parenting Intervention for Substance-Abusing Mothers. Psychoanal Psychol. 2008 Jul 1;25(3):499-517. doi: 10.1037/0736-9735.25.3.499. PMID 20057923
- [Result] Suchman, N., DeCoste, & Mayes, L. (2009). The Mothers and Toddlers Program: An attachment-based intervention for mothers in substance abuse treatment. In C. Zeanah (Ed.), Handbook of infant mental health, 3rd edition, pp. 485-499. New York, NY: Guilford Press.
- [Result] Suchman NE, DeCoste C, Castiglioni N, McMahon TJ, Rounsaville B, Mayes L. The Mothers and Toddlers Program, an attachment-based parenting intervention for substance using women: post-treatment results from a randomized clinical pilot. Attach Hum Dev. 2010 Sep;12(5):483-504. doi: 10.1080/14616734.2010.501983. PMID 20730641
- [Result] Suchman NE, Decoste C, McMahon TJ, Rounsaville B, Mayes L. THE MOTHERS AND TODDLERS PROGRAM, AN ATTACHMENT-BASED PARENTING INTERVENTION FOR SUBSTANCE-USING WOMEN: RESULTS AT 6-WEEK FOLLOW-UP IN A RANDOMIZED CLINICAL PILOT. Infant Ment Health J. 2011 Jul;32(4):427-449. doi: 10.1002/imhj.20303. Epub 2011 Jun 14. PMID 22685361
- [Result] Suchman NE, DeCoste C, Leigh D, Borelli J. Reflective functioning in mothers with drug use disorders: implications for dyadic interactions with infants and toddlers. Attach Hum Dev. 2010 Nov;12(6):567-85. doi: 10.1080/14616734.2010.501988. PMID 20931415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All mothers enrolled in outpatient substance use treatment and caring for a child between birth and 36 months of age were eligible. Mothers were recruited via clinician referrals and self-referral. Mothers who were actively suicidal, homicidal, severely cognitively impaired, disengaged from their treatment or not fluent in English were excluded.
Pre-assignment Details: Mothers were informed that after completing a baseline assessment they would be randomly assigned to one of two parenting programs. Mothers were asked permission to access their clinic attendance records and urinary toxicity results over the course of the study.
Groups:
- Mentalizing Therapy for Mothers: This 12 session individual therapy aims to enhance maternal reflective functioning and soften harsh and distorted mental representations about the child. The intervention adopts a developmental progression based on attachment theory, supporting the mother in her parenting role and offering assistance with basic needs. Mothers are encouraged to reflect on their thoughts and feelings and how they affect behavior. The therapist assists mother's thinking about representations of herself as a parent and encourages her to explore opportunities for new understanding of her emotional needs. Therapist and mother explore representations of her child and their relationship in detail in order to understand their meaning and promote more balanced representations and affect regulation. Therapist and mother also explore child's emotional experiences underlying behavior. The goal is to support the mother in becoming more aware of her child's emotional needs.
- Standard Parent Education: This 12 session comparison intervention was designed to match the Maternal Mentalizing Therapy on time spent with the counselor and maternal expectations for help with parenting. PE counselors helped mothers get connected to services (e.g. medical and pediatric care, child care and child guidance services, housing assistance, vocational training), solve problems of daily living and make parenting-related decisions. PE mothers also received a pamphlet each week on a parenting topic of their choice. Pamphlets focused on common issues in caring for infants (e.g., soothing a crying baby, managing bedtime routines, and establishing routines ) and toddlers (e.g., helping toddlers dress, managing bedtime battles, managing difficult behavior in public, and setting limits without using punishment). Pamphlets provided behavioral guidance at a 5th grade reading level without reference to underlying mental states or emotional needs.
Period: Overall Study
Arm/Group | Mentalizing Therapy for Mothers | Standard Parent Education
Started | 23 | 24
Completed | 17 | 17
Not Completed | 6 | 7
Not completed — Withdrawal by Subject | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mentalizing Therapy for Mothers | Standard Parent Education | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.43 (6.46) | 28.88 (6.50) | 30.16 (6.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Maternal Capacity for Reflective Functioning (Assessed With the Parent Development Interview)
Description: The Parent Development Interview (PDI) was used to measure maternal capacity to mentalize about her own and her child's behavior. The PDI is a 1 hour semi-structured interview designed to elicit the mother's narrative about commonly occurring, emotionally-challenging aspects of parenting. A rating of 1 indicates a absence of recognition of mental states. A rating of 3 indicates a limited capacity to acknowledge mental states. A rating of 5 indicates the presence of a rudimentary capacity for reflective functioning.
Time Frame: post-treatment and 6-week follow up
Population: Data analysis was conducted for ITT sample. Baseline data was available for 47 mothers. Missing post-tx and follow up scores for mothers who left treatment early were estimated as equal to baseline scores. Post-tx and follow up scores for mothers who completed treatment but not post-tx or follow up visits were estimated as equal to tx group means.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentalizing Therapy for Mothers | Standard Parent Education
Number analyzed (Participants) | 23 | 24
units on a scale
  Mentalizing for Self at post-treatment | 3.59 (.65) | 3.08 (.65)
  Mentalizing about Child at post-treatment | 3.54 (.54) | 3.47 (.54)
  Mentalizing for Self at 6-week follow up | 3.47 (.59) | 3.09 (.59)
  Mentalizing about Child at 6-week follow up | 3.45 (.39) | 3.37 (.39)

2. Primary Outcome: Quality of Maternal Representations of the Child (Assessed With the Working Model of the Child Interview)
Description: The Working Model of the Child Interview (WMCI; Zeanah & Benoit, 1993) is a 1.5 hour interview used to elicit a narrative description of the mother's perceptions of her child and their relationship. The rater was trained to reliably code 6 qualitative subscales: Openness, Richness, Coherence, Caregiving Sensitivity and Acceptance and Involvement. On the mean of six subscales, a score of three is considered to represent average representational quality, scores of 1 and 2 are considered to represent clinical risk and scores of 4 and 5 are considered to represent optimal quality.
Time Frame: post-treatment, 6-week follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentalizing Therapy for Mothers | Standard Parent Education
Number analyzed (Participants) | 23 | 24
units on a scale
  Maternal Representations at post-treatment | 2.86 (.40) | 2.78 (.40)
  Maternal Representations at 6-wk follow up | 2.86 (.32) | 2.71 (.32)

3. Secondary Outcome: Maternal Caregiving Behavior (Assessed With the NCAST Teaching Scales)
Description: Mothers choose a task to teach the child in a 5 minute teaching session. Maternal behavior is coded on 4 dimensions: Sensitivity to Cues, Response to Distress, Social-Emotional Growth Fostering, & Cognitive Growth Fostering. The Total Caregiver Score is the sum of the 4 subscale scores (73 items) with scores ranging from 0 to 73. The Total Caregiver Contingency Score is the sum of 20 items from the 4 subscales that involve the caregiver's contingent response to child cues (scores range from 0 to 20). Higher score are better and lower scores are worse. For mothers with high school education (which a majority in our sample had) here are the normative means (SDs) reported in the scoring manual: Total Caregiver Score = 40.69 (6.85), Sensitivity to Cues = 9.16 (1.62), Response to Distress = 10.04 (1.78), Social-Emotional Growth = 8.99 (1.83), Cognitive Growth = 12.51 (3).
Time Frame: post-treatment, 6-week follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentalizing Therapy for Mothers | Standard Parent Education
Number analyzed (Participants) | 23 | 24
units on a scale
  Total Caregiver Score at post-treatment | 37.79 (3.45) | 35.75 (3.44)
  Total Caregiver Contingency Score at post-treatmen | 14.60 (1.93) | 13.01 (1.93)
  Total Caregiver Score at 6-wk follow up | 37.06 (3.39) | 34.61 (3.38)
  Total Caregiver Contingency Score at 6-wk follow u | 13.62 (1.73) | 12.14 (1.73)

4. Secondary Outcome: Child Behavior (Assessed With the NCAST Teaching Scales)
Description: Child behavior with the mother was assessed using the Clarity of Cues and the Responsiveness to Caregiver Subscales from the NCAST Teaching Scales. The Child Total Score is the sum of the 2 scales (23 items) with scores ranging from 0 to 23. The Child Contingency Score is the sum of 12 contingent items from the 2 scales (with scores ranging from 0 - 12). The 2 subscores are summed to arrive at the composite score. Higher scores are better. The normative means for the children of high school educated mothers reported in the scoring manual: Total Child Score = 15.44 (4.29), Clarity of Cues = 7.99 (1.49), Responsiveness to Parent = 7.45 (3.16).
Time Frame: post-treatment and 6-wk follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentalizing Therapy for Mothers | Standard Parent Education
Number analyzed (Participants) | 23 | 24
units on a scale
  Child Total Score at post-treatment | 19.74 (2.44) | 18.78 (2.43)
  Child Contingency Score at post-treatment | 9.47 (1.57) | 9.16 (1.56)
  Child Total Score at 6-wk follow up | 20.16 (2.12) | 18.66 (2.12)
  Child Contingency Score at 6-wk follow up | 9.61 (1.48) | 9.11 (1.47)

5. Secondary Outcome: Maternal Depression (Measured With the Beck Depression Inventory)
Description: The Beck Depression Inventory (BDI; Beck, Steer, & Brown, 1996) was used to assess maternal symptoms of depression. The BDI is a widely used 21-item questionnaire rated on a 4-point scale and yields a total score ranging from 0 to 63: scores between 13 and 19 indicate mild depression; scores between 20 and 28 indicate moderate levels of depression, and scores between 29 and 63 indicate severe levels of depression (Beck et al., 1996).
Time Frame: post-treatment and 6-wk follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentalizing Therapy for Mothers | Standard Parent Education
Number analyzed (Participants) | 23 | 24
units on a scale
  Maternal Depression at post-treatment | 13.57 (7.30) | 16.01 (7.28)
  Maternal Depression at 6-wk follow up | 14.37 (6.66) | 12.14 (6.65)

6. Secondary Outcome: Maternal Psychiatric Distress (Assessed With the Brief Symptom Inventory)
Description: The Brief Symptom Inventory (BSI; Derogatis, 1993) was used to assess maternal global psychiatric distress. The BSI is a standardized, widely used, 53-item, 5-point, self-report measure of psychopathology. The composite Global Severity Index (GSI) measures current overall symptomatology across multiple domains and has demonstrated good reliability and validityT-scores have a mean of 50 and a standard deviation of 10. Scores within one standard deviation (ie. a T-score of 10) above the mean on any dimension are regarded as being within the normal range on that dimension (Derogatis, 1993). These scores were converted to T-scores using data from the scoring manual. The higher the scores are worse.T scores above 60 on the GSI indicate risk for a clinical disorder.
Time Frame: post-treatment and 6-wk follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mentalizing Therapy for Mothers | Standard Parent Education
Number analyzed (Participants) | 23 | 24
units on a scale
  Maternal Psychiatric Distress at post-treatment | 58.86 (6.71) | 60.24 (6.71)
  Maternal Psychiatric Distress at 6-wk follow up | 58.41 (6.71) | 58.29 (6.71)

7. Secondary Outcome: Maternal Substance Abuse (Assessed With Urine Toxicology Screens)
Description: Maternal substance use was monitored weekly using results from weekly urine toxicology (UTOX) screens testing for presence of opiate, cocaine, and cannabis metabolites in urine samples collected at the outpatient clinic. For each month of the mother's participation in the study, a mother received a score of "0" if no drug metabolites were present in any of her urine toxicology screens during that month or a score of "1" if one or more of her urine toxicology screens tested positive for a drug metabolite during that month. A percentage was calculated by= number of positive substance tests/number of total test *100 for each patients during each month.
Time Frame: post-treatment and 6-wk follow up
Population: as for outcome 1
Measure: Mean (Standard Error); unit: % positive utox screens/month
Arm/Group | Mentalizing Therapy for Mothers | Standard Parent Education
Number analyzed (Participants) | 23 | 24
% positive utox screens/month
  Maternal Substance use at post-treatment | 20 (.36) | 22 (.36)
  Maternal Substance use at 6-wk follow up | 7 (.22) | 6 (.22)

ADVERSE EVENTS:
Arm/Group | Mentalizing Therapy for Mothers | Standard Parent Education
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

LIMITATIONS AND CAVEATS:
Sample most representative of addicted mothers in mid-30's, Caucasian, high school educated, unemployed, moderate involvement with child welfare. Caution in generalizing to higher risk mothers (adolescent mothers, ethnic minority,less educated).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No